CLINICAL TRIAL: NCT04992624
Title: Cannabinoid Interactions With Central and Peripheral Pain Mechanisms in Osteoarthritis of the Knee
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Steven E Harte, PhD (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Steven E Harte, PhD, Associate Professor of Anesthesiology and Internal Medicine Associate Director, Chronic Pain and Fatigue Research Center, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: HUM000180986; 1R01AT010381-01A1 (NIH); 1K01DA049219-01A1 (NIH)
Record Dates: First submitted 2021-07-28; First posted 2021-08-05 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis of the Knee
Keywords: Cannabidiol; Tetrahydrocannabinol
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Cannabidiol; Dronabinol

STUDY DESIGN:
Intervention Model Description: This is a single-site, 2x2 factorial double-blind, randomized clinical trial with 200 participants (160 completers).
Who Masked: Participant, Investigator
Masking Description: Some of the treatment phase will be blinded by the study team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Cannabidiol (CBD) (Experimental): Up to 150 mg/day.
  Interventions: Drug: Cannabidiol (CBD)
- Tetrahydrocannabinol (THC) (Experimental): Up to 10 mg/day.
  Interventions: Drug: Tetrahydrocannabinol (Marinol® or generic equivalent (e.g., dronabinol)
- CBD plus THC (Experimental): Up to 150 mg/day CBD plus up to 10 mg/day THC.
  Interventions: Drug: Cannabidiol (CBD); Drug: Tetrahydrocannabinol (Marinol® or generic equivalent (e.g., dronabinol)

INTERVENTIONS:
Drug: Placebo — Placebo drug will be taken similarly to the THC and CBD and be matched to keep the trial blinded.
  In the event that 2.5 mg capsules of dronabinal capsules become unavailable, an equivalent product will be issued to participants and the comparator and placebo arms will be correspondingly adjusted to preserve blinding. If a participant's dose is not well-tolerated, the participant may initiate dose reductions with the study team.
  Participants will be instructed to eat a meal or snack greater than one hour after taking study drug.
  Arms: Placebo
Drug: Cannabidiol (CBD) — Epidiolex doses will be 0.37 milliliter (mL) for seven days of treatment and then 0.75 mL two times a day (b.i.d) for the remaining days of this treatment.
  In the event that 2.5 mg capsules of dronabinal capsules become unavailable, an equivalent product will be issued to participants and the comparator and placebo arms will be correspondingly adjusted to preserve blinding. If a participant's dose is not well-tolerated, the participant may initiate dose reductions with the study team.
  Participants will be instructed to eat a meal or snack greater than one hour after taking study drug.
  Other Names: Epidiolex
  Arms: CBD plus THC; Cannabidiol (CBD)
Drug: Tetrahydrocannabinol (Marinol® or generic equivalent (e.g., dronabinol) — Dronabinol Capsules doses will be 2.5 mg b.i.d. for seven days of treatment and then 5 mg b.i.d. for the remaining days of this treatment.
  In the event that 2.5 mg capsules of dronabinal capsules become unavailable, an equivalent product will be issued to participants and the comparator and placebo arms will be correspondingly adjusted to preserve blinding. If a participant's dose is not well-tolerated, the participant may initiate dose reductions with the study team.
  Participants will be instructed to eat a meal or snack greater than one hour after taking study drug.
  Other Names: Dronabinol
  Arms: CBD plus THC; Tetrahydrocannabinol (THC)

SUMMARY:
This clinical trial is being done to better understand how daily treatment with Tetrahydrocannabinol (THC), Cannabidiol (CBD), or the combination of CBD plus THC affects knee osteoarthritis pain and other related symptoms.

Consented participants will have a screening period and visit (up to 30 days to treatment start). If participants pass the screening phase, they will be randomly assigned to take one of the investigational study drugs. For this study, participants will not know when or if they are taking CBD, THC, THC plus CBD, and when or if taking placebo.

Clinical pain will be assessed at multiple times throughout the study, and eligibility will be re-assessed at two weeks into the treatment period. It is possible that subjects will not be able to participate in the study after 14 days of of treatment. The treatment period will take approximately 16 weeks and then a follow-up period for approximately 2 weeks. In addition to treatment, participants will have clinical assessments, blood draws, questionnaires, daily pain diaries, sensory testing, as well as have functional connectivity magnetic resonance imaging (fcMRI).

DETAILED DESCRIPTION:
The study hypothesizes that:

* CBD alone will exert a peripheral anti-inflammatory effect by decreasing levels of Interleukin (IL)-6
* THC alone will modify central nervous system (CNS) pain via decreasing insula to Default Mode Network (DMN) connectivity
* CBD plus THC will do both.

ELIGIBILITY:
Inclusion Criteria:

* Ability to read and speak English to allow for written informed consent, phenotyping, and patient-reported outcomes measures
* Willingness to participate in a drug intervention trial
* Diagnosis of osteoarthritis (OA) of the knee by a medical provider (confirmed by checking medical records)
* Chronic knee pain, defined as moderate to severe knee pain for ≥ 6-month duration
* No use of cannabis or CBD in the past in the month prior to study enrollment as per self-report
* Fibromyalgia (FM) Survey Criteria score available. The questionnaire will be assessed by the research team for scoring. We will recruit enough patients to satisfy the spectrum of FM scores in four quartiles based on our previously existing data. Once a quartile is filled (approximately 40 patients enrolled), then we will not include more people from that quartile.
* Self-reported normal visual acuity or correctable (with corrective lenses- glasses or contacts) to at least 20/40 for reading instructions in the MRI and visual sensitivity testing
* No contraindications to magnetic resonance imaging (MRI) (for example (e.g.), metal implants)
* Able to lie still on their back for 1-1.5 hours during MRI
* Willingness to refrain from pain medications such as non-steroidal anti-inflammatory drugs (NSAIDs) and acetaminophen for 12 hours prior to neuroimaging and Quantitative Sensory Testing (QST)
* Willingness to refrain from alcohol and nicotine before QST and neuroimaging (alcohol and nicotine consumption is allowed after testing is completed)
* Willingness to refrain from physical activity or exercise that would cause significant muscle and/or joint soreness for 48 hours prior to testing (routine exercise or activity that does not lead to soreness is acceptable)
* Willingness to maintain a stable treatment regimen for chronic knee OA pain during the clinical trial (e.g., not initiating a new course of physical therapy)
* No use of adjunctive pain medications or stable chronic daily use of adjunctive pain medications (excluding opioids)
* Willingness to avoid grapefruit juice or food products for the duration of the study;
* Females of reproductive potential must agree to use acceptable birth control from the screening visit and until the completion study drug administration. Sexually active male participants and/or their female partners must agree to use effective contraception during study drug treatment of the male participant. Male participants may also agree not to donate sperm during study drug treatment

Exclusion Criteria:

* Individuals who are actively applying for or in litigation for compensation or disability and other aspects associated with potential secondary gain per self-report
* Inability to provide written informed consent
* Previous total knee arthroplasty
* Planned total knee arthroplasty within the time frame of the study
* Severe physical impairment (e.g., blindness, deafness, paraplegia)
* Co-morbid medical conditions that may significantly impair physical functional status (e.g., history of non-skin malignancy, or autoimmune disorder)
* Use of cannabis or CBD in the past month per self-report and/or drug screen
* Current opioid use (excepting tramadol) per self-report and/or drug screen
* Current valproate, clobazam, or warfarin use per self-report or medical records
* Current use of moderate or strong inhibitors of cytochrome p450 (CYP) enzymes CYP3A4 and CYP2C19, strong inducers of CYP3A4 or CYP2C19, moderate or strong inhibitors/inducers of CYP2C9, and narrow therapeutic index drugs (e.g., cyclosporine, amphotericin B). Participants will also not be allowed to start using these drugs during the study period if they wish to stay in the study
* Self-reported allergies to sesame oil or cannabis/cannabinoids
* Self-reported medical or psychiatric conditions that in the judgment of study personnel would preclude participation in this study (e.g., schizophrenia, malignancy, psychosis, suicidal ideation, history of substance abuse; note that stable anxiety and depression are not exclusions)
* Pregnant or nursing
* Liver failure
* Self-reported liver cirrhosis
* Active diagnosis or current symptoms of hepatitis by self-report
* Self-reported uncontrolled diabetes
* Blood pressure at screening above 180 systolic and/or 120 diastolic
* Resting heart rate at screening less than 50 beats per minute (bpm) or greater than 100 bpm;
* Elevated liver enzymes and bilirubin (measured via blood test at screening):

  * Serum total bilirubin ≥ 2.5 milligrams per deciliter (mg/dL); or,
  * Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) ≥ 3x upper limit normal (ULN); or,
  * Alkaline phosphatase ≥ 2 times ULN
* Severe cardiovascular disease (examples: history of myocardial infarction, unstable angina, severe coronary artery disease, congestive heart failure, or severe valvular abnormalities) that is self-reported by patient or by medical record
* Severe claustrophobia precluding MRI
* Unable to fit in or lie comfortably in MRI
* Diagnosed peripheral neuropathy
* Diagnosed or self-reported epilepsy or history of seizures
* Current head injury or history of head injury (e.g., traumatic brain injury)
* Any impairment, activity, behavior, or situation that in the judgment of the study team would prevent satisfactory completion of the study protocol

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2026-10-22 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Default mode network (DMN) to insula connectivity via functional connectivity magnetic resonance imaging (fcMRI) | Day 15, and approximately day 99 of treatment
  Functional connectivity difference maps of insula to DMN connectivity using Independent Component Analysis and seed based connectivity. A reduction in the Z-score as a result of treatment will serve as the primary outcome measure.
Change in pre-post measurements of inflammatory marker IL-6. | Day 15, and approximately day 99 of treatment
  Serum IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Steve Harte, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No